CLINICAL TRIAL: NCT05572489
Title: Frequency of Cognitive Dysfunction in Individuals With Cervicogenic Headache
Brief Title: Cervicogenic Headache, Cognitive Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savaş Karpuz, Medical doctor, Konya Beyhekim Training and Research Hospital
Other Study IDs: 2021-01-02
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with cervicogenic headache: visual pain scale Beck depression scale Pain catastrophizing scale Short Form-36 Standard Mini mental test Montreal cognitive assessment scale
  Interventions: Diagnostic Test: visual pain scale Beck depression scale Pain catastrophizing scale Short Form-36 Standard Mini mental test Montreal cognitive assessment scale
- healthy controls: visual pain scale Beck depression scale Pain catastrophizing scale Short Form-36 Standard Mini mental test Montreal cognitive assessment scale
  Interventions: Diagnostic Test: visual pain scale Beck depression scale Pain catastrophizing scale Short Form-36 Standard Mini mental test Montreal cognitive assessment scale

INTERVENTIONS:
Diagnostic Test: visual pain scale Beck depression scale Pain catastrophizing scale Short Form-36 Standard Mini mental test Montreal cognitive assessment scale — evaluation of pain, fatigue, mood, quality of life, cognitive status

SUMMARY:
The goal of this study was to determine the frequency of cognitive dysfunction in patients with cervicogenic headache.

participants will be asked questions to determine their cognitive status at once.

DETAILED DESCRIPTION:
A set of survey-type questions will be asked to the participants. Pain and fatigue levels of the patients were measured by visual pain scale (VAS), mood states by Beck depression scale (BDI) and Pain catastrophizing scale (Pain catastrophizing scale), quality of life by Short Form-36 (SF-36), and cognitive status by Standard Mini. mental test (SMMT) and Montreal cognitive assessment scale (MOCA).

ELIGIBILITY:
Inclusion Criteria:

Clinical Diagnosis of cervicogenic headache be over 18

Exclusion Criteria:

those under the age of 18 Those with neurological deficits Those with rheumatic diseases such as fibromyalgia, polymyalgia rheumatica, ankylosing spondylitis, rheumatoid arthritis Surgery in the cervical region in the past 6 months Those with widespread pain, significant pain in another anatomical location (eg, gonarthrosis) Those who use drugs or substances (alcohol, drugs, etc.) that may cause cognitive impairment Those with known neurological diseases such as cerebrovascular disease, MS, Parkinson's, dementia Those with major psychiatric illness Those with communication problems Those who have started psychiatric medical treatment in the last three months Those with significant hearing or vision problems Those with a history of uncontrollable systemic disease (cardiovascular, pulmonary, hepatic, renal, hematological, endocrine..)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 30 patients with cervicogenic headache and 30 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
cognitive status | 01.12.2022

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Research and Training Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Shared on request.

REFERENCES:
- [Background] Bogduk N, Govind J. Cervicogenic headache: an assessment of the evidence on clinical diagnosis, invasive tests, and treatment. Lancet Neurol. 2009 Oct;8(10):959-68. doi: 10.1016/S1474-4422(09)70209-1. PMID 19747657
- [Background] Sjaastad O. Cervicogenic headache: comparison with migraine without aura; Vaga study. Cephalalgia. 2008 Jul;28 Suppl 1:18-20. doi: 10.1111/j.1468-2982.2008.01610.x. PMID 18494988